CLINICAL TRIAL: NCT01424254
Title: The Effectiveness of Video-capsule Endoscopy in Gastrointestinal Bleeding of Obscure Origin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); American College of Gastroenterology (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Alan Barkun, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: REC#03-025
Record Dates: First submitted 2011-08-18; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Gastrointestinal Bleeding
Keywords: Gastrointestinal Bleeding of Obscure Origin
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Double-Balloon Enteroscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video-Capsule Endoscopy (Experimental): VCE will be performed in the early morning following 200 mg of simethicone and 250 - 500 mg of erythromycin (as per physician's prescription), ingestion also in the absence of contra-indications
  Interventions: Device: Capsule GIVEN IMAGING
- Push Enterosopy (Experimental)
  Interventions: Procedure: Push-Enteroscopy

INTERVENTIONS:
Device: Capsule GIVEN IMAGING — Injection of Capsule Endoscopy
  Arms: Video-Capsule Endoscopy
Procedure: Push-Enteroscopy — currently recommended standard
  Arms: Push Enterosopy

SUMMARY:
The study objective is to compare the cost-effectiveness of VCE to push enteroscopy in patients with gastrointestinal bleeding of obscure origin with a negative initial work-up.

DETAILED DESCRIPTION:
Background: The introduction of the wireless capsule endoscopy (WCE) may dramatically alter the management of patients with small bowel disease such as chronic gastrointestinal bleeding of obscure origin (CGB). Yet, to date, this non invasive technique has undergone widespread diffusion in the absence of properly designed prospective comparative cost-effectiveness evaluations.

Objectives: To examine the clinical impact and cost-effectiveness of a novel approach employing WCE compared to that of push enteroscopy (PE).

Hypothesis: WCE is more cost-effective than PE in patients with CGB. Study design: We propose a randomized clinical trial comparing WCE to PE. Study population: Patients with CGB having undergone initial normal assessment with gastroscopy, colonoscopy and radiological examination of the small bowel.

Outcomes: Primary objective: To compare the detection rates of "clinically significant" small bowel lesions using WCE versus PE in CGB patients randomized to either modality. Secondary objectives: To determine the "cure rate" for each technique after 6 months, the cost-effectiveness of WCE versus PE, the type of small bowel lesions most likely to impact on clinical care, inter-rater variability in reading WCE examinations, the feasibility of WCE interpretation by a dedicated technician, the safety of each imaging modality, and to compare patient satisfaction and quality of life between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Normal gastroscopy, colonoscopy and small bowel follow through in the last 3 months

Exclusion Criteria:

* Demonstrable source of blood outside the GI tract
* Significant cardiopulmonary disease
* Suspicion of strictures or fistulae of the GI tract
* Pregnancy
* Numerous small intestinal diverticula
* Zenker's diverticulum
* Extensive Crohn's enteritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2003-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the detection rate of clinically significant lesions thought to be responsible for the patients with gastrointestinal bleeding of obscure origin | 12 months

SECONDARY OUTCOMES:
resolution of the anemia/recurrent bleeding | 12 months
blood transfusion requirements | 12 months
Number of required imaging tests (i.e: gastroscopy, colonoscopy, etc) | 12 months
hospitalization/length of stay | 12 months
days away from usual activities (protocol unrelated) | 12 months
patient satisfaction | Following procedure at randomization
  Patient satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada